CLINICAL TRIAL: NCT03042793
Title: Vaccination With PD-L1 Peptide With Montanide Against Multiple Myeloma After High Dose Chemotherapy With Stem Cell Support. A Phase I First-in-human Study.
Brief Title: Vaccination With PD-L1 Peptide Against Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lene Meldgaard Knudsen (Other)
Responsible Party: Sponsor-Investigator, Lene Meldgaard Knudsen, MD, DMSc, Head of Department, Department of Haematology, Universityhospital Herlev and Gentofte, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MY0001; 2016-000990-19 (EudraCT Number)
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Multiple Myeloma
Keywords: myeloma; vaccination; PD-L1; peptide vaccine; cancer vaccine; immunotherapy
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccination (Experimental): Vaccine: PD-L1 peptide.
  Interventions: Biological: PD-L1 peptide vaccine

INTERVENTIONS:
Biological: PD-L1 peptide vaccine — PD-L1 peptide given subcutaneously with Montanide ISA-51

SUMMARY:
Title: Vaccination with PD-L1 peptide with Montanide against multiple myeloma after high dose chemotherapy with stem cell support. A phase I first-in-human study.

Hypothesis: In this trial the investigators assess a new immunotherapeutic strategy targeting the immune checkpoint molecule PD-L1 to investigate the potential of vaccination against PD-L1 as a possible anticancer target.

DETAILED DESCRIPTION:
Background: Multiple myeloma is the second most common hematologic cancer which is despite advances in treatment is still incurable for most patients.

In this trial the investigators assess a new immunotherapeutic strategy targeting the immune checkpoint molecule PD-L1 to investigate the potential of vaccination against PD-L1 as a possible anticancer target.

PD-L1 has been recognized as an important factor in immune regulation and development of immune tolerance in the microenvironment of cancer cells. Cells that express PD-L1 on their surface are known to inhibit the immune system. As seen with the recent advances in immunotherapy against cancer with antibodies against PD-L1, the the immunosuppressive role of the molecule PD-L1 can be antagonized to the benefit of patients with cancer. PD-L1 is expressed on both cancer cells, antigen presenting cells and immunosuppressive cells in the tumor micro-environment. Vaccination against PD-L1 is therefore two sided. The investigators aim to stimulate PD-L1 specific T-cells, hence eliminating both PD-L1 positive tumor cells as well as PD-L1 positive immunosuppressive and antigen presenting cells in the tumor microenvironment. The primary endpoints are safety and toxicity evaluation. Secondary endpoint is immunological response. Clinical response will be described.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically verified multiple myeloma
2. Newly treated with HDT and no signs of relapse
3. Age ≥18 years
4. Performance status ≤ 2 (ECOG-scale)
5. Expected survival > 3 months
6. Sufficiently regenerated bone marrow function, i.e.

   1. Leucocytes ≥ 1,5 x 109
   2. Granulocytes ≥ 1,0 x 109
   3. Thrombocytes ≥ 20 x 109
7. Creatinine < 2.5 upper normal limit, i.e. < 300 μmol/l
8. Sufficient liver function, i.e.

   1. ALAT < 2.5 upper normal limit, i.e. ALAT <112 U/l
   2. Bilirubin < 30 U/l
9. Women agreement to use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 120 days after the last treatment.
10. For men: agreement to use contraceptive measures and agreement to refrain from donating sperm.

Exclusion Criteria:

1. Non-secretory myeloma
2. Other malignancies in the medical history excluding squamous cell carcinoma of the skin and patients cured for another malignant disease with no sign of relapse three years after ended treatment.
3. Significant medical condition per investigators judgement e.g. severe Asthma/COPD, poorly regulated heart condition, insulin dependent diabetes mellitus.
4. Acute or chronic viral infection e.g. HIV, hepatitis or tuberculosis
5. Serious known allergies or earlier anaphylactic reactions.
6. Known sensibility towards Montanide ISA-51
7. Any active autoimmune diseases e.g. autoimmune neutropenia, thrombocytopenia or hemolytic anemia, systemic lupus erythematosus, scleroderma, myasthenia gravis, autoimmune glomerulonephritis, autoimmune adrenal deficiency, autoimmune thyroiditis etc.
8. Pregnant and breastfeeding women.
9. Fertile women not using secure contraception with a failure rate less than < 1%
10. Patients taking immune suppressive medications incl. corticosteroids and methotrexate at the time of enrollment
11. Psychiatric disorders that per investigator judgment could influence compliance.
12. Treatment with other experimental drugs
13. Treatment with other anti-cancer drugs - except bisphosphonates and denosumab
14. Patients with active uncontrolled hypercalcemia
15. Patients who have received chemotherapy, immune therapy, radiation therapy within the last 28 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity | 12 months
  CTCAE = Common Terminology Criteria for Adverse Events v. 4.0 will be used for registration of toxicity

SECONDARY OUTCOMES:
Evaluation of immunological responses | 12 months
  Immunological assays will be used to identify immunological responses.

OTHER OUTCOMES:
Clinical response | 12 months
  Will be described according to standard IMWG-criteria for multiple myeloma.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Jørgensen, MD, Principal Investigator — Center for Cancer Immune Therapy, Universityhospital Herlev and Gentofte
Locations (1):
- Department of Hematology, Universityhospital Herlev and Gentofte, Herlev, Denmark

REFERENCES:
- [Derived] Jorgensen NG, Klausen U, Grauslund JH, Helleberg C, Aagaard TG, Do TH, Ahmad SM, Olsen LR, Klausen TW, Breinholt MF, Hansen M, Martinenaite E, Met O, Svane IM, Knudsen LM, Andersen MH. Peptide Vaccination Against PD-L1 With IO103 a Novel Immune Modulatory Vaccine in Multiple Myeloma: A Phase I First-in-Human Trial. Front Immunol. 2020 Nov 9;11:595035. doi: 10.3389/fimmu.2020.595035. eCollection 2020. PMID 33240282